CLINICAL TRIAL: NCT03069131
Title: A Multicenter, Double-blind, Placebo-controlled Randomized Clinical Trial Comparing Two Strategies of Primary Prophylaxis of Spontaneous Bacterial Peritonitis in Severe Cirrhotic Patients With Ascites : Using or Not Using Rifaximin
Brief Title: Two Strategies of Primary Prophylaxis of Spontaneous Bacterial Peritonitis in Severe Cirrhotic Patients With Ascites
Acronym: ProPILARifax
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Collaborators: Alfasigma S.p.A. (Industry); LC2 PHARMA (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ProPILA-Rifax
Record Dates: First submitted 2017-02-27; First posted 2017-03-03 (Actual); Last update posted 2025-04-10 (Actual); Status verified 2025-01

CONDITIONS: Cirrhosis; Ascites; Peritonitis
Keywords: primary prophylaxis; rifaximin
MeSH Terms: conditions — Fibrosis; Ascites; Peritonitis | interventions — Rifaximin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active rifaximin (Experimental)
  Interventions: Drug: Rifaximin
- Rifaximin placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Rifaximin — twice daily administration of 1 tablet containing 550 mg of active rifaximin
  Arms: Active rifaximin
Other: Placebo — twice daily administration of 1 rifaximin placebo tablet
  Arms: Rifaximin placebo

SUMMARY:
We wish to perform a multicenter, double-blind RCT with two parallel-group stratified on the center, comparing rifaximin to no rifaximin (placebo) for the primary prophylaxis of SBP in 'severe' cirrhotic patients with large ascites. The primary outcome will be the 12-month survival.

ELIGIBILITY:
Inclusion Criteria:

* Cirrhosis diagnosed on clinical, radiological and/or histological findings
* Patients with large ascites (i.e., grade 3 ascites requiring paracentesis). Patients with grade 2 ascites are also authorized.
* Ascites with a low protein level in ascitic fluid (< 15 g/L) with one of the following three conditions:

  1. impaired renal function defined by serum creatinine ≥ 106 mmol/L, uremia ≥ 9 mmol/L or serum sodium ≤ 130 mmol/L), or
  2. severe liver impairment defined by Child-Pugh score ≥ 9 with serum total bilirubin levels ≥ 51 mmol/L.
  3. severe liver impairment defined by Child-Pugh C
* Patient who signed an informed consent form
* Patient with a social security system
* Woman must be surgically sterile or be postmenopausal, or must agree to use effective contraception during the study if childbearing potential.
* Patients who needs a TIPS if the procedure is performed 3 months or more following the randomization
* Patients with severe alcoholic hepatitis can be considered for inclusion if the MELD score < 30 and the Maddrey Discriminant Function < 60 providing that the patient is not infected (and consequently, will not receive antibiotics) and has not yet received corticosteroid (if necessary). Patients not responding to corticosteroid at day 7 (according to the Lille score) could be include after a wash-out of steroids for a period of 7 days.

Exclusion Criteria:

* Pregnant woman or breastfeeding
* Vulnerable person regarding french law
* Individual under legal protection measure
* Individual unable to exprim his/her consent
* Person under 18 years of age and over 80 years of age
* Transplanted patients, HIV infection (or patients who deny HIV serology) or immunosuppressive therapy (including patients under corticosteroids for severe alcoholic hepatitis if the patients respond to steroids with improvement of liver function)
* Patients with a liver transplant project and an estimated waiting time for liver transplantation of 3 months or less
* Past SBP or any present bacterial infection
* Patient who have received a TIPS procedure before rhe randomization
* Patients with an alfapump
* Patient receiving antibiotics (including rifaximin) in the 7 days preceding the inclusion in this study exept for patients participating to the microbiota study (15 days).
* Hypersensitivity to rifaximin, derivatives of rifamycin or one of the constituents of the preparation
* Hepatocellular carcinoma outside the Milan criteria, other cancer at a palliative stage
* Any clinical situation with a very low short-terme prognosis (other than cirrhosis), i.e. a survival estimated lower than one month
* Gastrointestinal bleeding within 7 days
* Intestinal obstruction
* Grade 3 hepatic encephalopathy (HE) during the previous 6 months before randomization
* Chronic heart failure (stage III or IV of the New York Heart Association [NYHA] Functional Classification
* Patient judged as noncompliant
* Patients who cannot receive a clear information and who have no trusted relatives
* Patient who refuses the participation agreement by signing the information form and consent as defined in the protocol.
* Exclusion period from another biomedical study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2018-06-05 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2023-03-20 (Actual)

PRIMARY OUTCOMES:
death | 12 months
  record of death whatever the cause

SECONDARY OUTCOMES:
Hospital mortality rate and mortality rate at 3 months | 3 months
  survival during hospitalization and at 3 months
Hospital mortality rate and mortality rate at 6 months | 6 months
  survival during hospitalization and at 6 months
Incidence of spontaneous bacterial peritonitis (SBP) during follow-up | 12 months
  Bacterial analysis of ascites
Incidence of the other complications of liver cirrhosis during follow-up | 12 months
  complications of liver cirrhosis : SBP, HE, gastrointestinal bleeding and hepatorenal syndrome
Patient hospitalizations during follow-up | 12 months
  number of days of hospitalization during 12 months of follow-up
Quantitative variations of IL-6 in serum between day 1 and day 30 | 1 month
  Dosage of IL-6 in serum at D1 and D30
Quantitative variations of lipopolysaccharides (LPS) in serum between day 1 and day 30 | 1 month
  Dosage of LPS in serum at D1 and D30
Quantitative variations of copeptin in serum between day 1 and day 30 | 1 month
  Dosage of copeptin in serum at D1 and D30
Quantitative variations of CRP in serum between day 1 and day 30 | 1 month
  Dosage of CRP in serum at D1 and D30
Quantitative variations of von Willebrand Factor antigen in serum between day 1 and day 30 | 1 month
  Dosage of von Willebrand Factor antigen in serum at D1 and D30
Composition of the intestinal microbiota | up to 18 months
  analyzis of microbiota (quantity and quality of main bacterial strains) in 25 patients from arms A and B at day 1, and at months 3, 6, 12 and 18
Safety analysis of the study drug | 12 months
  Record of adverse events and serious adverse events in each arm

CONTACTS AND LOCATIONS:
Overall Officials: Rodolphe Anty, MD, Principal Investigator — Centre Hospitalier Universitaire de Nice; Edouard Bardou-Jacquet, MD, Principal Investigator — Rennes University Hospital; Christophe Bureau, MD, PhD, Principal Investigator — University Hospital, Toulouse; Vincent Di Martino, MD, PhD, Principal Investigator — CHRU de Besançon; Claire Francoz, MD, Principal Investigator — Hôpital Beaujon, Clichy; Alexandra Heurgue-Berlot, MD, Principal Investigator — CHU de Reims; Marianne Latournerie, MD, Principal Investigator — Centre Hospitalier Universitaire Dijon; Alexandre Louvet, MD, PhD, Principal Investigator — CHRU de Lille; Pierre Nahon, MD, PhD, Principal Investigator — Hôpital Jean Verdier, Bondy; Frédéric Oberti, MD, Principal Investigator — University Hospital, Angers; Isabelle Rosa-Hezode, MD, Principal Investigator — CHIC de Créteil; Marika Rudler, MD, Principal Investigator — Hôpital Pitié-Salpêtrière, APHP; Matthieu Schnee, MD, Principal Investigator — Hôpital La Roche-sur-Yon; Ghassan Riachi, MD, Principal Investigator — CHU Rouen; Isabelle Ollivier, MD, Principal Investigator — CHU CAEN; Eric Nguyen-Khac, MD, PhD, Principal Investigator — CHU Amiens; Laure Elkrief, MD, Principal Investigator — CHU Tours; Lucy Meunier, MD, Principal Investigator — University Hospital, Montpellier; Fanny Lebosse, MD, Principal Investigator — Hopital de la Croix-Rousse; Marie Noelle Hilleret, MD, Principal Investigator — University Hospital, Grenoble
Locations (18):
- France (18):
  - CHU Amiens, Amiens
  - CHU d'Angers, Angers
  - CHU de Besançon, Besançon
  - Hôpital Jean Verdier, Bondy
  - CHU Caen, Caen
  - Hôpital Beaujon, Clichy
  - CHIC de Créteil, Créteil
  - CHU Grenoble, La Tronche
  - CHRU de Lille, Lille
  - Hopital de la croix-rousse, Lyon
  - CHU Montpellier, Montpellier
  - CHU de Nice, Nice
  - Hôpital Pitié Salpêtrière, Paris
  - CHU de Reims, Reims
  - CHU de Rennes, Rennes
  - CHU Rouen, Rouen
  - CHU de Toulouse, Toulouse
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Thevenot T, Elkrief L, Bureau C, Bardou-Jacquet E, Rosa I, Nguyen-Khac E, Oberti F, Pitta A, Mallet M, Lebosse F, Louvet A, Meunier L, Nahon P, Ollivier-Hourmand I, Anty R, Francoz C, Riachi G, Meunier A, Cervoni JP, Tio G, Muller A, Cure-Martin A, Ladeira R, Clairet AL, Hocquet D, Di Martino V, Weil D, Desmarets M. Effect of rifaximin in patients with severe cirrhosis and ascites: A randomized double-blind placebo-controlled trial. J Hepatol. 2025 Dec;83(6):1320-1327. doi: 10.1016/j.jhep.2025.06.019. Epub 2025 Jul 11. PMID 40653111

DOCUMENTS (1):
  • Statistical Analysis Plan (2023-11-28): https://cdn.clinicaltrials.gov/large-docs/31/NCT03069131/SAP_001.pdf